CLINICAL TRIAL: NCT05764681
Title: Chronic Postsurgical Pain in Cerebral Palsy
Brief Title: Chronic Postsurgical Pain
Acronym: CPSP
Status: Recruiting | Type: Observational
Sponsor: Chantel Burkitt (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Minnesota (Other); Nemours Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Chantel Burkitt, Principal Investigator, Gillette Children's Specialty Healthcare
Organization: Gillette Children's Specialty Healthcare (Other)
Other Study IDs: STUDY00014668; 1R01HD108406-01A1 (NIH)
Record Dates: First submitted 2023-02-02; First posted 2023-03-13 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy; Chronic Post Surgical Pain
Keywords: Cerebral Palsy; Pain; Chronic Pain; Post Surgical Pain; Orthopedic Surgery
MeSH Terms: conditions — Cerebral Palsy; Pain, Postoperative; Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study purpose is to document the typical trajectory of perioperative pain experience in Cerebral Palsy (CP) and to identify important predictive factors for the development of chronic postsurgical pain. The main aims of the investigators are to:

1. Quantify the trajectory of pain and opioid use in the context of orthopedic surgery in children with CP.
2. Identify predictors for CPSP in children with CP and develop an applicable risk index.
3. Examine relationships between perioperative pain severity and functional/mobility outcomes achieved by orthopedic surgery in children with CP.

Participants will complete:

1. Questionnaires/Surveys via email and text message
2. In-person Sensory Tests
3. In-person Gait and Motion Analysis

ELIGIBILITY:
Inclusion Criteria:

* CP diagnosis
* Have a scheduled lower extremity or spine orthopedic surgery

Exclusion Criteria:

* Non-English speaking and reading parent/guardian

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Individuals with Cerebral Palsy undergoing an orthopedic surgery at Gillette Children's Specialty Healthcare or Nemour's Children Hospital, Delaware
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Change in Brief Pain Inventory (BPI) score from 1 week preoperative to 1, 3, 6, and 12 months postoperative | 1 month preoperative, and 1, 3, 6, and 12 months postoperative
  The BPI assesses pain location, pain intensity at worst, least, average, and right now as well as the degree to which pain interferes with activities of daily living (e.g., sleep, relationships, and mobility). Items are scored on an 11-point scale (0 = does not interfere, 10 = completely interferes) creating a total interference score ranging from 0-120 (higher scores mean more pain interference). The BPI has been adapted for and tested with individuals with severe CP, resulting in excellent internal consistency (Cronbach's alpha = 0.89) and validity evidence [1, 29, 30]. The BPI will take parents/children 1-2 minutes to complete.

SECONDARY OUTCOMES:
Dalhousie Pain Interview (DPI) | 1 month preoperative, and 1, 3, 6, and 12 months postoperative
  The DPI uses a 10-item survey to quantify pain intensity (Primary outcome variable; scored 0-10 with higher scores indicating more pain), duration (minutes/seconds in pain), and pain frequency (number of pain episodes) for each type of pain reported in the last week. The type and dose of pain-related medications is also collected. The DPI was developed to assess acute and chronic pain in children with developmental disabilities. The investigative team has considerable experience with the DPI and pain parameters have shown sensitivity to change after treatment [30, 31]. The DPI will take parents/children 5-15 minutes to complete.
Numeric Rating Scale (NRS) | From Post-Operative Day (POD) 3-90
  The NRS of pain is considered the 'gold standard' and has been widely used to quantify pain intensity (0-10 scale; 0=no pain, 10=worst possible pain). We will use the NRS specific to head, shoulders, upper arm, elbow, forearm, wrist/hand, back, hip, upper leg, knee, lower leg, ankle, and foot pain. The NRS will complement the DPI since it is joint-specific, which is a critical element to capture when assessing orthopedic outcomes. The NRS will take parents/children 3 minutes to complete.
SNAKE (Schlaffragebogen für Kinder mit Neurologischen und Anderen Komplexen Erkrankungen)Sleep Questionnaire | 1 month preoperative, and 1, 3, 6, and 12 months postoperative
  We will also collect the SNAKE Sleep Questionnaire via parent-report, a 43-item tool that measures the sleep environment, sleep patterns, and sleep behaviors (scores ranging from 23-92 with higher scores indicating more sleep difficulties). This tool was designed specifically for individuals with severe disabilities, and individuals with CP were included in the validation sample. The SNAKE will take parents 2-5 minutes to complete.
Gait Outcomes Assessment List (GOAL) | Any time preoperative and 12 months postoperative
  The GOAL had initial data published on it in 2011 [33]. It was developed for individuals with ambulatory CP and their parents as a comprehensive assessment of gait-related function. It is an outcome tool that incorporates all domains of the International Classification of Functioning, Disability and Health, including the influence of environment and personal factors [34].It contains 7 different domains and scores for each domain and for the total survey are standardized and range from 0 (worst) to 100 (best). A novel component of the GOAL is that it also incorporates the family's priorities for treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Chantel Burkitt, PhD, Principal Investigator — Gillette Children's, University of Minnesota
Locations (2):
- United States (2):
  - Nemour's Children's Hospital, Wilmington, Delaware
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barney CC, Stibb SM, Merbler AM, Summers RLS, Deshpande S, Krach LE, Symons FJ. Psychometric properties of the brief pain inventory modified for proxy report of pain interference in children with cerebral palsy with and without cognitive impairment. Pain Rep. 2018 Jul 17;3(4):e666. doi: 10.1097/PR9.0000000000000666. eCollection 2018 Jul-Aug. PMID 30123858
- [Background] Chidambaran V, Ding L, Moore DL, Spruance K, Cudilo EM, Pilipenko V, Hossain M, Sturm P, Kashikar-Zuck S, Martin LJ, Sadhasivam S. Predicting the pain continuum after adolescent idiopathic scoliosis surgery: A prospective cohort study. Eur J Pain. 2017 Aug;21(7):1252-1265. doi: 10.1002/ejp.1025. Epub 2017 Mar 27. PMID 28346762
- [Background] Delafontaine A, Presedo A, Mohamed D, Lopes D, Wood C, Alberti C. Equimolar mixture of nitroux oxyde and oxygen during post-operative physiotherapy in patients with cerebral palsy: A randomized, double-blind, placebo-controlled study. Eur J Pain. 2017 Nov;21(10):1657-1667. doi: 10.1002/ejp.1071. Epub 2017 Jul 20. PMID 28726270
- [Background] Boyer ER, Stout JL, Laine JC, Gutknecht SM, Araujo de Oliveira LH, Munger ME, Schwartz MH, Novacheck TF. Long-Term Outcomes of Distal Femoral Extension Osteotomy and Patellar Tendon Advancement in Individuals with Cerebral Palsy. J Bone Joint Surg Am. 2018 Jan 3;100(1):31-41. doi: 10.2106/JBJS.17.00480. PMID 29298258
- [Background] Dreher T, Thomason P, Svehlik M, Doderlein L, Wolf SI, Putz C, Uehlein O, Chia K, Steinwender G, Sangeux M, Graham HK. Long-term development of gait after multilevel surgery in children with cerebral palsy: a multicentre cohort study. Dev Med Child Neurol. 2018 Jan;60(1):88-93. doi: 10.1111/dmcn.13618. Epub 2017 Nov 24. PMID 29171016
- [Background] Munger ME, Aldahondo N, Krach LE, Novacheck TF, Schwartz MH. Long-term outcomes after selective dorsal rhizotomy: a retrospective matched cohort study. Dev Med Child Neurol. 2017 Nov;59(11):1196-1203. doi: 10.1111/dmcn.13500. Epub 2017 Aug 8. PMID 28786493
- [Background] Thomason P, Baker R, Dodd K, Taylor N, Selber P, Wolfe R, Graham HK. Single-event multilevel surgery in children with spastic diplegia: a pilot randomized controlled trial. J Bone Joint Surg Am. 2011 Mar 2;93(5):451-60. doi: 10.2106/JBJS.J.00410. PMID 21368077
- [Background] Wilson NC, Chong J, Mackey AH, Stott NS. Reported outcomes of lower limb orthopaedic surgery in children and adolescents with cerebral palsy: a mapping review. Dev Med Child Neurol. 2014 Sep;56(9):808-14. doi: 10.1111/dmcn.12431. Epub 2014 Mar 28. PMID 24673603
- [Background] Geil D, Thomas C, Zimmer A, Meissner W. Chronified Pain Following Operative Procedures. Dtsch Arztebl Int. 2019 Apr 12;116(15):261-266. doi: 10.3238/arztebl.2019.0261. PMID 31130157
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331
- [Background] Tucker A, McCusker D, Gupta N, Bunn J, Murnaghan M. Orthopaedic Enhanced Recovery Programme for Elective Hip and Knee Arthroplasty - Could a Regional Programme be Beneficial? Ulster Med J. 2016 May;85(2):86-91. PMID 27601761
- [Background] Totsch SK, Quinn TL, Strath LJ, McMeekin LJ, Cowell RM, Gower BA, Sorge RE. The impact of the Standard American Diet in rats: Effects on behavior, physiology and recovery from inflammatory injury. Scand J Pain. 2017 Oct;17:316-324. doi: 10.1016/j.sjpain.2017.08.009. Epub 2017 Sep 18. PMID 28927908
- [Background] Barney CC, Tervo R, Wilcox GL, Symons FJ. A Case-Controlled Investigation of Tactile Reactivity in Young Children With and Without Global Developmental Delay. Am J Intellect Dev Disabil. 2017 Sep;122(5):409-421. doi: 10.1352/1944-7558-122.5.409. PMID 28846038
- [Background] Barney CC, Merbler AM, Simone DA, Walk D, Symons FJ. Investigating the Feasibility of a Modified Quantitative Sensory Testing Approach to Profile Sensory Function and Predict Pain Outcomes Following Intrathecal Baclofen Implant Surgery in Cerebral Palsy. Pain Med. 2020 Jan 1;21(1):109-117. doi: 10.1093/pm/pnz114. PMID 31268147
- [Background] Haskett ME, Ahern LS, Ward CS, Allaire JC. Factor structure and validity of the parenting stress index-short form. J Clin Child Adolesc Psychol. 2006 Jun;35(2):302-12. doi: 10.1207/s15374424jccp3502_14. PMID 16597226
- [Background] Goubert L, Eccleston C, Vervoort T, Jordan A, Crombez G. Parental catastrophizing about their child's pain. The parent version of the Pain Catastrophizing Scale (PCS-P): a preliminary validation. Pain. 2006 Aug;123(3):254-263. doi: 10.1016/j.pain.2006.02.035. Epub 2006 Apr 27. PMID 16644128
- [Background] Engel JM, Wilson S, Tran ST, Jensen MP, Ciol MA. Pain catastrophizing in youths with physical disabilities and chronic pain. J Pediatr Psychol. 2013 Mar;38(2):192-201. doi: 10.1093/jpepsy/jss103. Epub 2012 Oct 1. PMID 23033363
- [Background] Breau LM, MacLaren J, McGrath PJ, Camfield CS, Finley GA. Caregivers' beliefs regarding pain in children with cognitive impairment: relation between pain sensation and reaction increases with severity of impairment. Clin J Pain. 2003 Nov-Dec;19(6):335-44. doi: 10.1097/00002508-200311000-00001. PMID 14600533
- [Background] Bursch B, Tsao JC, Meldrum M, Zeltzer LK. Preliminary validation of a self-efficacy scale for child functioning despite chronic pain (child and parent versions). Pain. 2006 Nov;125(1-2):35-42. doi: 10.1016/j.pain.2006.04.026. Epub 2006 Jun 5. PMID 16740360
- [Background] Duckworth AL, Quinn PD. Development and validation of the short grit scale (grit-s). J Pers Assess. 2009 Mar;91(2):166-74. doi: 10.1080/00223890802634290. PMID 19205937
- [Background] Perpina-Galvan J, Richart-Martinez M, Cabanero-Martinez MJ, Martinez-Dura I. Content validity of the short version of the subscale of the State-Trait Anxiety Inventory (STAI). Rev Lat Am Enfermagem. 2011 Jul-Aug;19(4):882-7. doi: 10.1590/s0104-11692011000400005. English, Portuguese, Spanish. PMID 21876939
- [Background] Connelly M, Fulmer RD, Prohaska J, Anson L, Dryer L, Thomas V, Ariagno JE, Price N, Schwend R. Predictors of postoperative pain trajectories in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2014 Feb 1;39(3):E174-81. doi: 10.1097/BRS.0000000000000099. PMID 24173016
- [Background] Fernandez-Blazquez MA, Avila-Villanueva M, Lopez-Pina JA, Zea-Sevilla MA, Frades-Payo B. Psychometric properties of a new short version of the State-Trait Anxiety Inventory (STAI) for the assessment of anxiety in the elderly. Neurologia. 2015 Jul-Aug;30(6):352-8. doi: 10.1016/j.nrl.2013.12.015. Epub 2014 Jan 28. English, Spanish. PMID 24484757
- [Background] Hermann C, Hohmeister J, Zohsel K, Ebinger F, Flor H. The assessment of pain coping and pain-related cognitions in children and adolescents: current methods and further development. J Pain. 2007 Oct;8(10):802-13. doi: 10.1016/j.jpain.2007.05.010. Epub 2007 Jul 12. PMID 17631054
- [Background] Ravens-Sieberer U, Gosch A, Rajmil L, Erhart M, Bruil J, Duer W, Auquier P, Power M, Abel T, Czemy L, Mazur J, Czimbalmos A, Tountas Y, Hagquist C, Kilroe J, Kidscreen Group E. KIDSCREEN-52 quality-of-life measure for children and adolescents. Expert Rev Pharmacoecon Outcomes Res. 2005 Jun;5(3):353-64. doi: 10.1586/14737167.5.3.353. PMID 19807604
- [Background] Hidecker MJ, Paneth N, Rosenbaum PL, Kent RD, Lillie J, Eulenberg JB, Chester K Jr, Johnson B, Michalsen L, Evatt M, Taylor K. Developing and validating the Communication Function Classification System for individuals with cerebral palsy. Dev Med Child Neurol. 2011 Aug;53(8):704-10. doi: 10.1111/j.1469-8749.2011.03996.x. Epub 2011 Jun 27. PMID 21707596
- [Background] Harrison, P.L., Oakland, T., Adaptive Behavior Assessment System, Third Edition [Manual]. 2015, Torrance, CA: Western Psychological Services.
- [Background] Bell KL, Benfer KA, Ware RS, Patrao TA, Garvey JJ, Arvedson JC, Boyd RN, Davies PSW, Weir KA. Development and validation of a screening tool for feeding/swallowing difficulties and undernutrition in children with cerebral palsy. Dev Med Child Neurol. 2019 Oct;61(10):1175-1181. doi: 10.1111/dmcn.14220. Epub 2019 Apr 1. PMID 30937885
- [Background] Breau LM, Camfield CS, McGrath PJ, Finley GA. The incidence of pain in children with severe cognitive impairments. Arch Pediatr Adolesc Med. 2003 Dec;157(12):1219-26. doi: 10.1001/archpedi.157.12.1219. PMID 14662579
- [Background] Barney CC, Krach LE, Rivard PF, Belew JL, Symons FJ. Motor function predicts parent-reported musculoskeletal pain in children with cerebral palsy. Pain Res Manag. 2013 Nov-Dec;18(6):323-7. doi: 10.1155/2013/813867. PMID 24308022
- [Background] Rivard PF, Nugent AC, Symons FJ. Parent-proxy ratings of pain before and after botulinum toxin type A treatment for children with spasticity and cerebral palsy. Clin J Pain. 2009 Jun;25(5):413-7. doi: 10.1097/AJP.0b013e31819a6d07. PMID 19454875
- [Background] Tyler EJ, Jensen MP, Engel JM, Schwartz L. The reliability and validity of pain interference measures in persons with cerebral palsy. Arch Phys Med Rehabil. 2002 Feb;83(2):236-9. doi: 10.1053/apmr.2002.27466. PMID 11833028
- [Background] Savedra MC, Holzemer WL, Tesler MD, Wilkie DJ. Assessment of postoperation pain in children and adolescents using the adolescent pediatric pain tool. Nurs Res. 1993 Jan-Feb;42(1):5-9. PMID 8424069
- [Background] Matson JL, Malone CJ. Validity of the sleep subscale of the Diagnostic Assessment for the Severely Handicapped-II (DASH-II). Res Dev Disabil. 2006 Jan-Feb;27(1):85-92. doi: 10.1016/j.ridd.2005.03.001. Epub 2005 May 31. PMID 15927446
- [Background] Blankenburg M, Tietze AL, Hechler T, Hirschfeld G, Michel E, Koh M, Zernikow B. Snake: the development and validation of a questionnaire on sleep disturbances in children with severe psychomotor impairment. Sleep Med. 2013 Apr;14(4):339-51. doi: 10.1016/j.sleep.2012.12.008. Epub 2013 Mar 1. PMID 23453904
- [Background] Jenkins BN, Kain ZN, Kaplan SH, Stevenson RS, Mayes LC, Guadarrama J, Fortier MA. Revisiting a measure of child postoperative recovery: development of the Post Hospitalization Behavior Questionnaire for Ambulatory Surgery. Paediatr Anaesth. 2015 Jul;25(7):738-45. doi: 10.1111/pan.12678. Epub 2015 May 9. PMID 25958978